CLINICAL TRIAL: NCT04287491
Title: Use Of Virtual Reality For Pain Control in Dermatological Bedside Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190653
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Group (Experimental): This group will receive the virtual reality intervention during out-patient bedside procedures.
  Interventions: Other: Oculus Go Virtual Reality System

INTERVENTIONS:
Other: Oculus Go Virtual Reality System — The VR system will provide a 3D environment that provides distracting stimulus. Participant will put on the Oculus Go VR system headset 1-2 minutes prior to out-patient bedside procedure up to the completion of procedure which takes typically 3-5 minutes.

SUMMARY:
The purpose of this research study is to explore the impact of virtual reality (VR) on pain perception during out-patient procedures such as wart removal, wound debridement, and lidocaine injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients 13 years and older.
* Patient (or health care proxy when applicable) must sign an ICF.
* Patient requiring any painful dermatological bedside procedure including: wound debridement, injections and liquid nitrogen application.
* Patients willing to participate and parents able to consent.

Exclusion Criteria:

* Subjects with a diagnosis of vertigo, inner ear diseases or seizures are excluded due to the uncertainty of performance under VR conditions.
* Subjects requiring procedures on the head are also excluded to the interference of the VR headset.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in average pain as assessed by the visual analog scale (VAS) | Baseline, up to 2 hours
  VAS has a scoring range from 0 to 10 with 0 being no pain and 10 being the worst possible pain.
Change in maximum pain level as assessed by VAS | Baseline, up to 2 hours
  VAS has a scoring range from 0 to 10 with 0 being no pain and 10 being the worst possible pain.

SECONDARY OUTCOMES:
Change in heart rate | Baseline, up to 2 hours
  Heart rate will be assessed in beats per minute.
Change in oxygen saturation | Baseline, up to 2 hours
  Oxygen saturation will be assessed as a percentage.
Incidence of intervention related adverse events | Baseline, up to 2 hours
  Intervention related adverse events will be assessed per treating physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No